CLINICAL TRIAL: NCT06659744
Title: Emulation of Effects of Injectable Semaglutide on Cardiovascular Outcomes in Individuals With Type 2 Diabetes: SUSTAIN6 Trial
Brief Title: Emulation of the SUSTAIN6 Diabetes Trial Using Healthcare Claims
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Associate Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2018P002966-DUP-SUSTAIN
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- New use of semaglutide injection: Exposure group
  Interventions: Drug: New use of semaglutide injection
- New initiation of sitagliptin: Reference group
  Interventions: Drug: New initiation of sitagliptin

INTERVENTIONS:
Drug: New use of semaglutide injection — New use of semaglutide injection dispensing claim is used as the exposure.
  Groups: New use of semaglutide injection
Drug: New initiation of sitagliptin — New initiation of sitagliptin dispensing claim is used as the reference.
  Groups: New initiation of sitagliptin

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale emulation of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the RCT DUPLICATE initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to emulate, as closely as is possible in healthcare insurance claims data, the trial listed below/above. Although many features of the trial cannot be directly emulated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization is also not emulable in healthcare claims data but was proxied through a statistical balancing of measured covariates according to standard practice. Investigators assume that the RCT provides the reference standard treatment effect estimate and that failure to replicate RCT findings is indicative of the inadequacy of the healthcare claims data for emulation for a range of possible reasons and does not provide information on the validity of the original RCT finding.

The SUSTAIN6 trial, is a non-inferiority trial to evaluate the effects of injectable semaglutide versus placebo in terms of cardiovascular safety (CV death, nonfatal MI, or nonfatal stroke) in patients with type 2 diabetes.

The database study designed to emulate SUSTAIN6 trial will be a new-user active comparative study, where we compare the effect of injectable semaglutide versus sitagliptin on MACE outcome among patients with T2DM. Sitagliptin was selected to act as an active-comparator proxy for placebo. Sitagliptin and the class of dipeptidyl peptidase-4 (DPP-4) inhibitors have been demonstrated not to have an effect on MACE in a series of RCTs, and they are used in similar stages of disease/line of therapy as semaglutide, as well as being of similar cost.

ELIGIBILITY:
Eligible cohort entry dates:

Market availability of injectable semaglutide in the US began on 5th December 2017.

Optum: Study period between 5th Dec 2017 - 29th February 2024 Marketscan: Study period between 5th Dec 2017 - 31st Dec 2022 Medicare: Study period between 5th Dec 2017 - 31st Dec 2020

Inclusion Criteria:

* Type 2 diabetes mellitus
* Anti-diabetic drug naïve, or treated with one or two oral antidiabetic drug (OADs), or treated with human Neutral Protamin Hagedorn (NPH) insulin or long-acting insulin analogue or pre-mixed insulin, both types of insulin either alone or in combination with one or two OADs
* Age above or equal to 50 years at screening and clinical evidence of cardiovascular disease: prior myocardial infarction, prior stroke or prior transient ischemic attack, prior coronary, carotid or peripheral arterial revascularization, more than 50% stenosis on angiography or imaging of coronary, carotid or lower extremities arteries, chronic heart failure - New York Heart Association (NYHA) class II-III, chronic renal impairment documents by estimated eGFR <60ml/min/1.73 m2 per MDRD
* Age 60 years or older with subclinical evidence of cardiovascular disease. Subclinical cardiovascular risk factors as one of the following: persistent microalbuminuria (30-299mg/g) or proteinuria, ankle/brachial index less than 0.9

Exclusion Criteria:

* Type 1 diabetes mellitus, secondary or gestational diabetes
* Use of glucagon-like peptide-1 (GLP-1) receptor agonist (exenatide, liraglutide, or other) or pramlintide within 90 days prior to screening
* Use of any dipeptidyl peptidase 4 (DPP-IV) inhibitor within 30 days prior to screening
* Treatment with insulin other than basal and pre-mixed insulin within 90 days prior to screening - except for short-term use in connection with intercurrent illness
* Acute decompensation of glycaemic control requiring immediate intensification of treatment to prevent acute complications of diabetes (eg diabetes ketoacidosis) within 90 days prior to screening
* History of chronic pancreatitis or idiopathic acute pancreatitis
* Acute coronary or cerebro-vascular event within 90 days prior to randomization
* Chronic heart failure New York Heart Association (NYHA) class IV
* Personal or family history of multiple endocrine neoplasia type 2 (MEN2) or familial medullary thyroid carcinoma
* Personal history of non-familial medullary thyroid carcinoma
* Chronic hemodialysis or peritoneal dialysis
* End stage liver disease
* A prior solid organ transplant or awaiting solid organ transplant
* Diagnosis of malignant neoplasm in the previous 5 years
* Female of childbearing potential who is pregnant, breast-feeding or intends to become pregnant or is not using an adequate contraceptive method
* Known use of non-prescribed narcotics or illicit drugs
* Proliferative retinopathy or maculopathy requiring treatment
* Missing age or gender
* Nursing home admission

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population included patients with Type 2 Diabetes (Type2DM) who had not been treated with antihyperglycemic agents or had been treated with no more than two oral antihyperglycemic agents, with or without NPH or long-acting insulin, >=50 years with established cardiovascular disease OR >=60 years with subclinical cardiovascular disease.
Sampling Method: Non-Probability Sample
Enrollment: 158310 (Actual)
Dates: Start 2024-10-24 (Actual); Primary Completion 2025-03-06 (Actual); Study Completion 2025-03-06 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac event (MACE), including myocardial infarction, stroke, and all cause death | Through study completion (1 day after cohort entry date until the first of outcome or censoring)
  Hazard ratio

OTHER OUTCOMES:
Cataract surgery (negative control) | Through study completion (1 day after cohort entry date until the first of outcome or censoring)
  Hazard ratio

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Kruger N, Schneeweiss S, Desai RJ, Sreedhara SK, Kehoe AR, Fuse K, Hahn G, Schunkert H, Wang SV. Cardiovascular outcomes of semaglutide and tirzepatide for patients with type 2 diabetes in clinical practice. Nat Med. 2025 Nov 9. doi: 10.1038/s41591-025-04102-x. Online ahead of print. PMID 41207920

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: Study Protocol for Three-Stage Project (2025-07-30): https://cdn.clinicaltrials.gov/large-docs/44/NCT06659744/Prot_SAP_004.pdf
  • Study Protocol and Statistical Analysis Plan: Study Protocol for Two-Stage Project (2025-04-23): https://cdn.clinicaltrials.gov/large-docs/44/NCT06659744/Prot_SAP_002.pdf
  • Study Protocol and Statistical Analysis Plan: Amendment to Study Protocol for Two-Stage Project (2025-10-05): https://cdn.clinicaltrials.gov/large-docs/44/NCT06659744/Prot_SAP_005.pdf